CLINICAL TRIAL: NCT02544594
Title: Randomized Clinical Study of Extra-Corporal Life Support in Cardiogenic Shock Complicating Acute Myocardial Infarction
Brief Title: Clinical Study of Extra-Corporal Life Support in Cardiogenic Shock Complicating Acute Myocardial Infarction
Acronym: ECLS-SHOCK
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: LMU Klinikum (Other)
Responsible Party: Principal Investigator, PD Dr. Stefan Brunner, PD Dr. med., LMU Klinikum
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GE IDE MucM001-15
Record Dates: First submitted 2015-09-02; First posted 2015-09-09 (Estimated); Last update posted 2019-10-14 (Actual); Status verified 2019-10

CONDITIONS: Cardiogenic Shock
MeSH Terms: conditions — Shock, Cardiogenic

STUDY DESIGN:
Intervention Model Description: Best medical therapy versus best medical therapy + ECLS in the treatment of cardiogenic shock complicating acute myocardial infarction
Oversight: Data Monitoring Committee: No

ARMS (2):
- Extra-Corporal Life Support (ECLS) (Active Comparator): Standard treatment plus Extra-Corporal Life Support (ECLS) (from Sorin) in patients with cardiogenic shock due to myocardial infarction.
  Interventions: Device: Extra-Corporal Life Support (ECLS)
- Standard treatment (No Intervention): Standard treatment alone without Extra-Corporal Life Support (ECLS) in patients with cardiogenic shock due to myocardial infarction.

INTERVENTIONS:
Device: Extra-Corporal Life Support (ECLS) — Extra-Corporal Life Support (ECLS) (from Sorin)
  Arms: Extra-Corporal Life Support (ECLS)

SUMMARY:
This study compares standard treatment plus Extra-Corporal Life Support (ECLS) versus standard treatment alone in patients with cardiogenic shock due to myocardial infarction.

DETAILED DESCRIPTION:
Cardiogenic shock is a serious complication of a myocardial infarction. Despite optimal treatment the mortality in patients with cardiogenic shock still exceeds 50% and surviving patients mostly suffer from severe heart failure due to an impaired cardiac function.

This study compares standard treatment plus Extra-Corporal Life Support (ECLS) versus standard treatment alone in patients with cardiogenic shock due to myocardial infarction.

The main study hypothesis is to explore if additional treatment with ECLS preserves cardiac function (left ventricular ejection fraction) in patients with cardiogenic shock complicating acute myocardial infarction.

ELIGIBILITY:
Inclusion Criteria:

Cardiogenic shock complicating acute myocardial (STEMI or NSTEMI) with

* intended revascularization (PCI or CABG)
* Systolic blood pressure < 90 mmHg > 30 min or inotropes required to maintain pressure > 90 mmHg during systole
* Signs of left heart insufficiency and pulmonary congestion
* Signs of impaired organ perfusion with at least one of the following:

  * Altered mental status
  * Cold, clammy skin
  * Urine output <30 ml/h
  * Serum lactate >2mmol/l
* Informed consent

Exclusion Criteria:

* Resuscitation > 60 minutes, ischemia > 10 minutes
* No intrinsic heart action
* Cerebral deficit with fixed dilated pupils
* Mechanical infarction complication
* Onset of shock > 12 h
* Severe peripheral artery disease
* Aortic regurgitation > II.°
* Age > 80 years
* shock of other cause
* Other severe concomitant disease
* participation in another trial

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2015-11; Primary Completion 2018-03 (Actual); Study Completion 2019-03 (Actual)

PRIMARY OUTCOMES:
Left ventricular ejection fraction (LVEF) on day 30 | 30 days

SECONDARY OUTCOMES:
30-day mortality | 30 days
Lactate levels | up to 48 hours
potentia hydrogenic levels | 48 hours
Length of mechanical ventilation | 30 days
Long-term mortality at 12 months | up to 12 months
Length of ICU stay | 30 days
Neurological Outcome (modified Rankin Scale) | up to 12 months
MACE (defined as cardiac death, non-fatal myocardial re-infarction, rehospitalisation for cardiac reasons and the need of CABG or PCI) | up to 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Brunner, MD, Principal Investigator — Munich University Hospital; Steffen Massberg, MD, Study Chair — Munich University Hospital
Locations (1):
- University Hospital Munich, Munich, Bavaria, Germany

REFERENCES:
- [Derived] Brunner S, Guenther SPW, Lackermair K, Peterss S, Orban M, Boulesteix AL, Michel S, Hausleiter J, Massberg S, Hagl C. Extracorporeal Life Support in Cardiogenic Shock Complicating Acute Myocardial Infarction. J Am Coll Cardiol. 2019 May 14;73(18):2355-2357. doi: 10.1016/j.jacc.2019.02.044. No abstract available. PMID 31072581